CLINICAL TRIAL: NCT07276867
Title: Intrathecal Dexmedetomidine-Fentanyl Combination Versus Fentanyl Alone as Adjuvant to Bupivacaine in Spinal Anesthesia for Above Knee Amputation in Sarcomas of Lower Extremity: A Randomized, Comparative Study
Brief Title: Intrathecal Dexmedetomidine-Fentanyl Combination Versus Fentanyl Alone as Adjuvant to Bupivacaine in Spinal Anesthesia for Above Knee Amputation in Sarcomas of Lower Extremity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mai Mohamed El Rawas, Assistant professor of Anaesthesia, Intensive Care and Pain Management, National Cancer Institute, Cairo University Cairo University, Cairo, Egypt., National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2509-501-125-203
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Intrathecal; Dexmedetomidine; Fentanyl; Bupivacaine; Spinal Anesthesia; Above Knee Amputation; Sarcomas; Lower Extremity
MeSH Terms: conditions — Sarcoma | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DF (Experimental): Patients will receive 2.5 mL of 0.5% hyperbaric bupivacaine with 25 µg fentanyl + 5 µg dexmedetomidine.
  Interventions: Drug: Fentanyl + Dexmedetomidine
- Group F (Active Comparator): Patients will receive 2.5 mL of 0.5% hyperbaric bupivacaine with 25 µg fentanyl.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl + Dexmedetomidine — Patients will receive 2.5 mL of 0.5% hyperbaric bupivacaine with 25 µg fentanyl + 5 µg dexmedetomidine.
  Arms: Group DF
Drug: Fentanyl — Patients will receive 2.5 mL of 0.5% hyperbaric bupivacaine with 25 µg fentanyl.
  Arms: Group F

SUMMARY:
The current work evaluated whether the combination of intrathecal dexmedetomidine and fentanyl provides superior postoperative analgesia to fentanyl alone when administered with hyperbaric bupivacaine.

DETAILED DESCRIPTION:
Above-knee amputation (AKA) for advanced lower limb (LL) sarcomas has a high risk of chronic pain syndromes, like phantom limb pain, and is associated with severe perioperative pain. Effective analgesia is essential for patient comfort, early rehabilitation, and improved outcomes.

Dexmedetomidine (DEX), a highly selective α2-adrenergic agonist, is a promising intrathecal (IT) adjuvant.

The combination of DEX and fentanyl may produce synergistic effects, extending block duration and improving perioperative analgesia while minimizing individual drug doses. The current approach is particularly relevant in oncologic surgeries like AKA, where optimal pain control is critical. However, supportive evidence exists in various surgical contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 60 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status of II-III.
* Height between 150-185 cm.
* Body mass index between 18-35 kg/m².
* Scheduled for above-knee amputation due to lower limb sarcomas.

Exclusion Criteria:

* Allergy to any of the investigated drugs.
* History of heart block, arrhythmia, or ongoing therapy with beta- or calcium channel- blockers, or angiotensin-converting-enzyme inhibitors.
* Contraindications to spinal anesthesia.
* Pregnancy or lactation.
* Presence of psychiatric illness or chronic pain conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 24 hours postoperatively
  Time to first rescue analgesia (time from the end of surgery till the first dose of morphine is administered).

SECONDARY OUTCOMES:
Total amount of morphine | 24 hours postoperatively
  If the Visual Analogue Scale (VAS) exceeded 3, rescue analgesia (RA) will be administered with intravenous morphine 3 mg.
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 0.5 µg/kg IV will be administered if heart rate or mean arterial blood pressure is elevated more than 20% of the baseline (after exclusion of other causes than pain).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at the Post-Anesthesia Care Unit (PACU), 2, 4, 6, 12, 18, and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as Nausea and vomiting, shivering, bradycardia, hypotension, and respiratory depression were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.